CLINICAL TRIAL: NCT06080568
Title: Energy Balance and Mitochondrial Function in Human Genetic Models of Mitochondrial Stress-mediated Obesity Resistance
Brief Title: Human Mitochondrial Stress-driven Obesity Resistance
Acronym: MITO-OB-RES
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Matteo Fiorenza, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: MITO-OB-RES
Record Dates: First submitted 2023-09-29; First posted 2023-10-12 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Mitochondrial Diseases; Mitochondrial Myopathies; Mitochondrial Disorder
Keywords: Energy balance; Energy expenditure; Appetite; Energy intake; Mitochondrial dysfunction
MeSH Terms: conditions — Mitochondrial Diseases; Mitochondrial Myopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, muscle tissue, subcutaneous adipose tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mitochondrial myopathy: Individuals with pathogenic mtDNA mutations
- Control: Individuals without mtDNA mutations

SUMMARY:
The overarching aim of this observational study is to determine alterations in energy balance while exploring the underlying cellular mechanisms in human genetic models of mitochondrial stress.

In a case-control design, individuals with pathogenic mitochondrial DNA mutations will be compared to healthy controls matched for sex, age, and physical activity level. Participants will attend a screening visit and an experimental trial including assessments of energy expenditure, appetite sensation, energy intake, and muscle and subcutaneous adipose tissue biopsy samples.

DETAILED DESCRIPTION:
Background: Pre-clinical models of mitochondrial stress are resistant to diet-induced obesity. Likewise, humans with primary mitochondrial diseases present a high prevalence of underweight (42%) as compared to a very low prevalence of obesity (2%). In this direction, recent data show a lower BMI across 17 cohorts of patients with mitochondrial diseases compared to national averages, suggesting mitochondrial stress-induced increments in resting energy expenditure as the primary driver of the lean phenotype. In recent years, the study of humans with genetic mutations has shown enormous potential to establish the mechanistic link between two physiological variables; indeed, if the mutation has a functional impact on one of those variables, then the direction of causality can be readily ascribed. Taken together, studies integrating assessments of energy balance with mitochondrial phenotyping in patients with rare mitochondrial disorders hold the potential to uncover putative mechanisms conferring protection from obesity in humans.

Objective: To determine alterations in energy expenditure/intake while exploring the underlying cellular mechanisms in individuals harboring mitochondrial DNA (mtDNA) mutations associated with mitochondrial stress.

Study design: Case-control study in individuals with mtDNA mutations (n=15) and healthy controls (n=15) matched for sex, age, and physical activity level.

Endpoint: Differences between individuals with mtDNA mutations and controls.

ELIGIBILITY:
Eligibility criteria for individuals with mitochondrial DNA mutations

Inclusion criteria:

- Known mtDNA point mutations

Exclusion criteria:

* Use of antiarrhythmic medications or other medications which, in the opinion of the investigators, have the potential to affect outcome measures.
* Diagnosed severe heart disease, dysregulated thyroid gland conditions, or other dysregulated endocrinopathies, or other conditions which, in the opinion of the investigators, have the potential to affect outcome measures.
* Pregnancy

Eligibility criteria for controls

Exclusion criteria:

* Current and regular use of antidiabetic medications or other medications which, in the opinion of the investigators, have the potential to affect outcome measures.
* Diagnosed heart disease, symptomatic asthma, liver cirrhosis or -failure, chronic kidney disease, dysregulated thyroid gland conditions or other dysregulated endocrinopathies, or other conditions which, in the opinion of the investigators, have the potential to affect outcome measures
* Daily use of tobacco products
* Excessive alcohol consumption
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with mitochondrial myopathy due to pathogenic mtDNA mutations are identified and recruited from the Copenhagen Neuromuscular Center or the Department of Clinical Genetics (Rigshospitalet).
  Control volunteers are recruited via recruitment announcements in Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Resting energy expenditure | Before (baseline) and 60-180 minutes after ingestion of a glucose solution
  Resting energy expenditure is measured in the fasting and fed state by indirect calorimetry
Appetite | Before (baseline) and 60-180 minutes after ingestion of a glucose solution as well as immediately after an ad libitum meal test
  Subjective appetite sensations are measured in the fasting and fed state by visual analogue scale (VAS) ratings
Energy intake | 180 minutes after ingestion of a glucose solution
  Energy intake is measured by quantifying the amount of food ingested during an ad libitum meal test

SECONDARY OUTCOMES:
Plasma hormones and cytokines modulating appetite and energy expenditure | Before (baseline) and 0-180 minutes after ingestion of a glucose solution
  Plasma levels of FGF21, GDF15, GLP-1, PYY, ghrelin, glucagon, and GIP are measured in the fasting and fed state
Plasma adipokines modulating appetite and energy expenditure | Baseline
  Plasma levels of leptin and adiponectin are measured in the fasting state
Muscle mitochondrial leak respiration | Baseline
  Mitochondrial O2 flux is measured by high-resolution respirometry in permeabilized muscle fibers
Muscle mitochondrial efficiency | Baseline
  Mitochondrial P/O ratio is measured by high-resolution respirometry in isolated mitochondria
Muscle mitochondrial membrane potential | Baseline
  Mitochondrial membrane potential is measured by high-resolution fluorometry in isolated mitochondria

OTHER OUTCOMES:
Body composition | Baseline
  Fat free mass and fat mass are determined by dual-energy X-ray absorptiometry
Physical activity level | Baseline
  Physical activity level is measured by wrist-worn accelerometers
Self-reported physical activity | Baseline
  Self-reported physical activity is measured by the International Physical Activity Questionnaire - Short Form (IPAQ-SF)
Cardiorespiratory fitness | Baseline
  Pulmonary maximal oxygen uptake (VO2max) is determined during an incremental exercise test to exhaustion

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Fiorenza, Ph.D., Principal Investigator — Rigshospitalet, Denmark; John Vissing, MD, Principal Investigator — Rigshospitalet, Denmark; Signe Torekov, Ph.D., Principal Investigator — University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo Q, Xu Z, Zhou D, Fu T, Wang W, Sun W, Xiao L, Liu L, Ding C, Yin Y, Zhou Z, Sun Z, Zhu Y, Zhou W, Jia Y, Xue J, Chen Y, Chen XW, Piao HL, Lu B, Gan Z. Mitochondrial proteostasis stress in muscle drives a long-range protective response to alleviate dietary obesity independently of ATF4. Sci Adv. 2022 Jul 29;8(30):eabo0340. doi: 10.1126/sciadv.abo0340. Epub 2022 Jul 27. PMID 35895846
- [Background] Yang M, Xu L, Xu C, Cui Y, Jiang S, Dong J, Liao L. The Mutations and Clinical Variability in Maternally Inherited Diabetes and Deafness: An Analysis of 161 Patients. Front Endocrinol (Lausanne). 2021 Nov 25;12:728043. doi: 10.3389/fendo.2021.728043. eCollection 2021. PMID 34899594
- [Background] Sturm G, Karan KR, Monzel AS, Santhanam B, Taivassalo T, Bris C, Ware SA, Cross M, Towheed A, Higgins-Chen A, McManus MJ, Cardenas A, Lin J, Epel ES, Rahman S, Vissing J, Grassi B, Levine M, Horvath S, Haller RG, Lenaers G, Wallace DC, St-Onge MP, Tavazoie S, Procaccio V, Kaufman BA, Seifert EL, Hirano M, Picard M. OxPhos defects cause hypermetabolism and reduce lifespan in cells and in patients with mitochondrial diseases. Commun Biol. 2023 Jan 12;6(1):22. doi: 10.1038/s42003-022-04303-x. PMID 36635485
- [Background] O'Rahilly S. "Treasure Your Exceptions"-Studying Human Extreme Phenotypes to Illuminate Metabolic Health and Disease: The 2019 Banting Medal for Scientific Achievement Lecture. Diabetes. 2021 Jan;70(1):29-38. doi: 10.2337/dbi19-0037. PMID 33355307
- [Background] Saleheen D, Natarajan P, Armean IM, Zhao W, Rasheed A, Khetarpal SA, Won HH, Karczewski KJ, O'Donnell-Luria AH, Samocha KE, Weisburd B, Gupta N, Zaidi M, Samuel M, Imran A, Abbas S, Majeed F, Ishaq M, Akhtar S, Trindade K, Mucksavage M, Qamar N, Zaman KS, Yaqoob Z, Saghir T, Rizvi SNH, Memon A, Hayyat Mallick N, Ishaq M, Rasheed SZ, Memon FU, Mahmood K, Ahmed N, Do R, Krauss RM, MacArthur DG, Gabriel S, Lander ES, Daly MJ, Frossard P, Danesh J, Rader DJ, Kathiresan S. Human knockouts and phenotypic analysis in a cohort with a high rate of consanguinity. Nature. 2017 Apr 12;544(7649):235-239. doi: 10.1038/nature22034. PMID 28406212